CLINICAL TRIAL: NCT03580629
Title: Pilot Study of the Liver Live Donor Champion Program
Acronym: LLDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00170784
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: End Stage Liver Disease
Keywords: Live Donor Liver Transplant; Education; Advocacy; Live Donor Champion
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Live Donor Champion (Experimental): The Liver Live Donor Champion program (LLDC) is the sole educational intervention for this trial. LLDC consists of 2 or 3 monthly sessions (depending on cohort) of approximately 2 or 3 hours each. Each LLDC session is led by a transplant physician or clinical coordinator. The sessions incorporate formal didactics, active-participant learning, personal stories, moderated group discussions, role-playing, and other skill-building exercises. LLDC session topics are as follows: 1) education about End-Stage Liver Disease (ESLD), liver transplantation, and living donation 2) communication skills building 3) Exploring social networks 4) sharing successful donor and recipient stories 5) surgeon and hepatologist panel 6) Program Recap.
  Interventions: Behavioral: Liver Live Donor Champion Program

INTERVENTIONS:
Behavioral: Liver Live Donor Champion Program — Even with adequate education of live donation, many liver transplant candidates still feel ill equipped to ask others to consider donating. Friends and family are often eager to help and may not be able to serve as donors themselves, but might be able to provide instrumental support. A Live Donor Champion (LDC) is a friend or family member who serves as an advocate for the candidate in their pursuit of live donation. The Johns Hopkins Comprehensive Transplant Center has developed the Liver Live Donor Champion program to provide education and advocacy training to waitlist candidates and their LDCs. The support provided by the LDC bridges a critical link between education and action. Using LDCs to increase live donation is a novel approach that has garnered widespread enthusiasm.
  Other Names: LLDC program

SUMMARY:
In this pilot study, investigators plan to enroll liver transplant candidates and a "Live Donor Champion" for an abridged two- or three-month program that provides education and advocacy training in order to expand access to live donor liver transplantation. Investigators have created two versions of the same program and based on feedback from participants and staff, investigators aim to analyze the efficacy of the Liver Liver Donor Champion program on this patient population.

DETAILED DESCRIPTION:
In the United States, more than 13,000 patients are on the waiting list to receive a liver transplant. Although more than 6,000 liver transplants are performed every year, at least 1,700 patients die each year while on the waiting list. Livers are allocated to patients based on how sick the participants are, with sicker patients receiving priority.

Living donation offers patients the option of transplant before patients get very sick, significantly decreasing the time patients wait for a liver. Livers from living donors are usually of excellent quality because donors are evaluated extensively and only allowed to donate if patients are in very good health. Living donation not only saves the life of the liver transplant candidate but also frees up a liver for a patient on the waiting list who does not have that option.

A number of studies have attempted to understand barriers to finding a living donor. Multiple surveys have suggested that the educational needs are not met for both transplant candidates and potential donors. Furthermore, lack of knowledge and understanding of the consequences of donation may aggravate candidate fear of donor risks, contributing to candidate reluctance in allowing friends or family to donate. Finally, having an inadequate communication skill set in how to ask someone to donate is one of the most prevalent barriers reported by transplant candidates.

A "Live Donor Champion" (LDC) is a friend, family member, or community member who serves as an advocate for the candidate in participants' pursuit of living donation. Investigators' center has previously developed a six-month program that provides education and advocacy training to kidney transplant candidates and participants' LDCs; however, no program currently exists for liver transplant candidates.

The instrumental support provided by the LDC from investigators' kidney program bridges a critical link between education and action. In pilot studies, candidates with an LDC were more likely to undergo live donor kidney transplantation than matched controls.

In this pilot study, investigators plan to enroll liver transplant candidates and participants' LDCs for an abridged two- or three-month program that provides education and advocacy training in order to expand access to live donor liver transplantation. Investigators have created two versions of the same program and based on feedback from participants and staff, investigators aim to analyze the efficacy of the Liver Liver Donor Champion program on this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Active candidate on the liver transplant waitlist.
* Have no potential living donors at the time of study enrollment.
* Have not had a previous transplant
* be 18 years or older
* be English speaking
* Mentally capable of providing informed consent

Exclusion Criteria:

* Age less than 18 years old
* Has potential live donor candidates
* non-English speaking
* Previous liver transplant
* Listed for multiple organs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-29 (Actual)

PRIMARY OUTCOMES:
Live Donor Inquiries | within 2 year of enrollment
  Live Donor Inquiries on behalf of candidates will be collected/identified through electronic medical system.
Live Donor Liver Transplantation | within 2 year of enrollment
  Live Donor Liver Transplantation within one year of enrollment into the study will be collected/identified through electronic medical record system.

SECONDARY OUTCOMES:
Knowledge of live donation and liver transplantation | within 6 months of enrollment
  Knowledge of live donation and liver transplantation will be collected during participant surveys.
Comfort initiating conversations | within 6 months of enrollment
  Comfort initiating conversations with others about live donation will be collected during participant surveys.
Feasibility - Implementation Outcome | within 2 year of enrollment
  Feasibility is defined as the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Feasibility will be assessed qualitatively by recording reflections of the implementing study team.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A King, MD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No